CLINICAL TRIAL: NCT06828640
Title: Treatment of Vulvo-vaginal Atrophy (VVA) Using Vaginal Dilator in Addition to Usual Treatment : a Randomized Control Trial
Brief Title: Treatment of Vulvo-vaginal Atrophy (VVA) Using Vaginal Dilator in Addition to Usual Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B0762024240710
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-08

CONDITIONS: Vulvo Vaginal Atrophy; Genitourinary Syndrome of Menopause (GSM); Vaginal Atrophy in Breast Cancer Patients; Vaginal Atrophy Patients With GSM; Treatment; Sexual Disfunction; Dyspareunia (Female)
Keywords: Vulvo vaginal atrophy; vaginal dilators; Genitourinary syndrome of menopause; treatment
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Intervention Model Description: Monocentric pilot RCT evaluating SoC (MHT, lubricants, moisturizers) (control group) to SoC + vaginal dilators (test group).
  SoC = Standard of care RCT = randomized control trial MHT = Menopausal hormonal therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group : vaginal dilators (Experimental): A Test group receiving the standard treatment + a kit of vaginal dilators with progressively larger sizes.
  Interventions: Device: vaginal dilators
- Control Group : placebo (No Intervention): A control group receiving the standard treatment (which includes MHT, vaginal lubricants, and Moisturizers).

INTERVENTIONS:
Device: vaginal dilators — Evaluate the efficacy of vaginal dilators as an addition to Standard of Care in premenopausal or menopausal women, including breast cancer survivors
  Arms: Test Group : vaginal dilators

SUMMARY:
This is a randomized, controlled trial aiming to evaluate the effectiveness of adding vaginal dilators to the treatment of vulvovaginal atrophy.

Study Population:

Peri- and postmenopausal women with VVA, including breast cancer survivors.

Design: Monocentric pilot RCT evaluating SoC (MHT, lubricants, moisturizers) (control group) to SoC + vaginal dilators (test group).

Vaginal Dilator : A silicone medical device will be used for gradual stretching progression. The kit includes dilators of progressively larger sizes.

Procedures: Assessments at baseline, at 4 & 12 weeks

Measures : Vulvo Vaginal Atrophy severity , dyspareunia, Vaginal Health Index Score, Female Sexual Fonction Index, and Visual Analogue Scale (for vaginal dryness, vaginal and/or vulvar irritation/itching, and pain during sexual intercourse).

Statistical Analysis:

Differences at baseline, 4 weeks, and 12 weeks will be tested using:

Two-sample t-test Mann-Whitney test

Statistical Power:

Assuming a 20% improvement in Group 1 and 40% in Group 2, with:

p < 0.05 (type I error) 80% power (type II error), 160 patients needed across both groups.

SoC = Standard of care RCT = Randimized control trial MHT = Menopausal hormonal therapy

ELIGIBILITY:
Inclusion Criteria:

* Peri- or postmenopausal women suffering from vulvovaginal atrophy (VVA)
* Breast cancer survivors with VVA symptoms
* Understand the study, be willing to participate, and sign an informed consent form.
* The use of estrogen/progestogen-based products (vaginal, oral, pellets, transdermal, etc.) is permitted but must be documented (this will be considered during randomization).

Exclusion Criteria:

* Undiagnosed abnormal genital bleeding.
* Administration of any investigational drug within 30 days prior to the screening visit.
* Presence of a serious medical condition, neurological disorder, or significant comorbidities.
* Other gynecological malignancies.
* Recent vaginal surgery.
* Clinically significant prolapse (POP-Q ≤ 2).
* Current urinary tract or vaginal infection, or recent sexually transmitted infection.
* Individuals with disabilities unable to communicate.
* Women eligible for the study but unwilling to participate.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
• Vaginal dryness score | At baseline, 4 and 12 weeks
  * None: no feeling of dryness.
  * Mild: occasional feeling of dryness that does not interfere with daily activities.
  * Moderate: feeling dry most of the time but does not interfere with daily activities.
  * Severe: continuous feeling of dryness interfering with daily activities.
• Vaginal and/or vulvar irritation/itching | At baseline, 4 and 12 weeks
  * None: no feeling of irritation.
  * Mild: occasional irritating sensation that does not interfere with daily activities.
  * Moderate: feeling irritated most of the time but does not interfere with daily activities.
  * Severe: continuous feeling of irritation interfering with daily activities.
• Pain during sexual intercourse score | At baseline, 4 and 12 weeks
  * None: pleasant sexual intercourse, rare pain.
  * Mild: occasional pain, not during every sexual intercourse, intercourse should be interrupted occasionally.
  * Moderate: most of the time, little satisfaction during intercourse and it often has to be interrupted.
  * Severe: during each sexual intercourse, no pleasure during intercourse and these must often be interrupted. Often post-coital bleeding. Frequent abstinence due to pain.
Vaginal Health index score | at baseline and 12 weeks
  The vaginal health score (VHIS) consists of analyzing five vaginal parameters: Vaginal elasticity; Volume of vaginal secretions; vaginal pH; the integrity of the epithelium of the vaginal walls and the lubrication/hydration of the vagina.
  For each vaginal parameter we give a score ranging from 1 to 5 The VHIS score is obtained by adding all the scores obtained (minimum score = 5 and maximum score = 25.
  If VHIS <15, the vagina is considered atrophic.
Patient satisfaction : visual analogue scale | At baseline, 4 and 12 weeks
  Evaluation of symptoms linked to vaginal atrophy (dryness, irritation, dyspareunia) on a visual analogue scale for pain (0 to 10) 0 = symptoms absent 10 = unbearable symptoms
Quality of life questionnaire specific to genitourinary syndrome | At baseline, 4 and 12 weeks
  Answer yes or no :
  Over the past week, have you been bothered by:
  Itchy vulva? Burning or tingling in the vulva? Pain in the vulva? Irritations to the vulva? Dryness in the vulva? Unpleasant vulvar or vaginal discharge? Odors coming from your vulva or vagina? Are you worried about your vulvar symptoms? (for example, will it spread, get worse, leave scars? etc.) Frustrations about your vulvar symptoms? Embarrassment about your vulvar symptoms? How do your vulvar symptoms affect your interactions with others? How do your vulvar symptoms affect your desire to be with people? Do your vulvar symptoms prevent you from showing affection? How do your vulvar symptoms affect your daily activities? Do your vulvar symptoms prevent you from having intimate relationships? The effects of your vulvar symptoms on your sexual relations? Do your vulvar symptoms cause pain during sexual activity? Do your vulvar symptoms cause dryness during sexual activity?
Female Sexual Function Index (FSFI) questionnaire | At baseline, 4 and 12 weeks
  * Desire Question :1, 2 Score range (1 - 5 ) min score 1.2 max score 6.0
  * Arousal Question : 3, 4, 5, 6 Score range( 0 - 5) min score : 0 Max score : 6.0
  * Lubrication: Question 7, 8, 9, 10 Score range(0 - 5) min score : 0 max score : 6.0
  * Orgasm : Question 11, 12, 13 Score range (0 - 5) min score 0 max score : 6.0
  * Satisfaction: Question : 14, 15, 16 Score range (0 (or 1) - 5) min score : 0.8 max score : 6.0
  * Pain : Question : 17, 18, 19 Score range(0 - 5) min score : 0 max score : 6.0
  Full Scale Score Range minimum score : 2.0 maximum score : 36.0

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | At 4 and 12 weeks
  Did you experience any side effects or discomfort related to the procedure?
  * Yes
  * No
    → If yes, can you specify which ones? 8. Have you considered stopping the procedure at any point?
  * Yes
  * No
Rate of adherence to the study by patients | At 4 and 12 weeks
  Was the intervention compatible with your lifestyle?
  * Yes, absolutely
  * Rather yes
  * Rather no
  * No, not at all 10. Did you encounter any obstacles in following the intervention?
  * Yes
  * No → If yes, can you specify which ones?

CONTACTS AND LOCATIONS:
Overall Officials: Serge Rozenberg, Gynaecologist, Study Director — Saint Pierre University Hospital Center
Locations (1):
- Saint Pierre University Hospital Center, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: October 2024 -2025 : 1 year
Access Criteria: on request

REFERENCES:
- [Background] Kingsberg SA, Wysocki S, Magnus L, Krychman ML. Vulvar and vaginal atrophy in postmenopausal women: findings from the REVIVE (REal Women's VIews of Treatment Options for Menopausal Vaginal ChangEs) survey. J Sex Med. 2013 Jul;10(7):1790-9. doi: 10.1111/jsm.12190. Epub 2013 May 16. PMID 23679050